CLINICAL TRIAL: NCT03489928
Title: A Randomized Controlled Trial of Oral Misoprostol, Low Dose Vaginal Misoprostol and Vaginal Dinoprostone for Induction of Labour
Brief Title: Misoprostol Labour Induction Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: David Young (Other)
Responsible Party: Sponsor-Investigator, David Young, Active Staff Physician, IWK Health Centre
Organization: IWK Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB#1415; 051.731.7303088 (Other Grant/Funding Number: IWK Research Services Grant)
Record Dates: First submitted 2018-03-06; First posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Induction of Labour; Labour, Induced
Keywords: Labour; Induction; Misoprostol; Dinoprostone; Oxytocin
MeSH Terms: interventions — Misoprostol; Dinoprostone; KLK15 protein, human

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of three approaches to initiation of labour induction. Study group allocation will be stratified based on membrane status (ruptured/intact). Sequentially numbered opaque envelopes contain group assignment prepared using computer generated random number tables, in blocks of 4 and 6. Group 1 will receive misoprostol 50µgs, repeated at 4hr intervals until one of the following occurs: progressive labour, contraction frequency of 3 per 10 minutes, non-reassuring fetal heart rate tracing, or delivery. Group 2 will receive misoprostol 25µg initial dose and then 25-50µg placed in the vagina at 6hr intervals to the same effect. Group 3 will have induction of labour managed by the usual method here at the IWK (intravaginal or intracervical prostaglandin gel and IV oxytocin drip). All care decisions will be made by the attending physician. The patient will be reassessed before each administration of misoprostol.
Masking Description: Group assignment will be concealed until time induction is to begin, when randomization will occur. No attempt will be made at formal blinding of caregivers following concealed randomization, although neonatal assessment will be carried out by a team unaware of study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Misoprostol (Experimental): 50ug po q4h orally, as needed
  Interventions: Drug: Oral Misoprostol
- Low dose vaginal misoprostol (Experimental): 25-50ug q6h, vaginally, as needed
  Interventions: Drug: Vaginal Misoprostol
- Usual vaginal dinoprostone (Experimental): 1-2mg q6h, vaginally as needed
  Interventions: Drug: Dinoprostone

INTERVENTIONS:
Drug: Oral Misoprostol — Prostaglandin E1 - 100ug tablet, divided in half by pharmacy staff to be administered by mouth.
  Other Names: Oral Cytotec
  Arms: Oral Misoprostol
Drug: Vaginal Misoprostol — Prostaglandin E1 - 100ug oral tablet, divided in quarters by pharmacy staff, vaginal placement of one or two quarters as needed every 6 hours
  Other Names: Vaginal Cytotec
  Arms: Low dose vaginal misoprostol
Drug: Dinoprostone — Prostaglandin E2 - 1-2mg gel manufactured for vaginal use; placed vaginally every 6 hours as needed.
  Other Names: Prostin
  Arms: Usual vaginal dinoprostone

SUMMARY:
Labour induction is a frequent obstetric intervention (~20%). Prostaglandins (PGs) are effective agents, but gastrointestinal (GI) intolerance has limited use to non-oral routes. The traditional oxytocin "drip" requires intravenous (IV) use and discourages mobility. Misoprostol, a PG analogue, is marketed for oral treatment of GI disorders, but initiates uterine contraction, an undesirable GI side effect. Recently, there has been a research "boom" on vaginal misoprostol use in pregnancy to induce term labour drawing on this "side effect:". The principal investigator has led one of three groups worldwide which has published on oral misoprostol to study effectiveness, GI tolerance, and safety for mother/baby in term labour induction. Cost per patient has been less then one percent that of other PGs, even less than IV oxytocin.

DETAILED DESCRIPTION:
Labour induction is a frequent obstetric intervention (20-30%). Prostaglandins (PGs) are effective agents, but gastrointestinal (GI) intolerance has limited use to intracervical and vaginal administration of PGE2 gels. Misoprostol, a prostaglandin E2 (PGE1) analogue, is marketed for oral treatment of upper GI disorders. The past five years has seen mushrooming literature on its use to initiate uterine contractions for pregnancy termination in the first and second trimesters, and labour induction in the third. Vaginal administration has been used almost exclusively, has been cost effective (less than one percent the cost of PGE2) and without demonstrated harm to mother or newborn. The investigators have published a randomized control trial (RCT) on vaginal use, and have also published a 275 subject RCT of oral misoprostol versus a traditional induction regime of (physician chosen combinations of intracervical or vaginal dinoprostone, intravenous (IV) oxytocin and artificial membrane rupture). Oral misoprostol was effective, well tolerated and without harm to mother or newborn. The investigators have in press a double blind RCT or oral versus vaginal misoprostol in 206 subjects. Oral misoprostol was effective, though time to vaginal birth was 226 min longer, due to more time before labour was initiated. Oral misoprostol was associated with less uterine hyperstimulation (P<0.04). The investigators have also completed an RCT of oral misoprostol versus IV oxytocin with term pre-labour membrane rupture. Again, effectiveness was shown. There is no larger published collective experience with oral misoprostol labour induction. Before embarking on a costly RCT to evaluate more substantive outcomes (Caesareans or neonatal asphyxia) with sample size greater than 10,000, funding has been received for this three-group RCT of labour induction at term: oral misoprostol, vaginal misoprostol, and our centre's established approach.

PRIMARY RESEARCH QUESTION When induction of labour at term is indicated, is there more than a four-hour difference in time to vaginal birth between vaginal misoprostol (25µg initial dose, followed by 25-50µg every six hours as needed), oral misoprostol (50µg every four hours as needed) and the Izaak Walton Killam (IWK) Health Centre established protocol? Secondary outcomes address harm to the newborn (including cord blood acid base analysis, and defined birth asphyxia criteria) and mother (Caesareans, peripartum interventions, maternal GI intolerance and excessive uterine activity).

RESEARCH PLAN Eligible subjects will be at gestations greater than 37 completed weeks, with a cephalic presenting live single fetus, who have an indication for induction, and no contraindication to induction, vaginal birth, or PG use. Random allocation will be blocked and stratified (on membrane status). Sample size calculations were based on: ∆=240 minutes, α(2 tailed) = 0.05, β=0.05, with a σ=588 minutes from the investigators' prior publications. Adjustments for anticipated Caesareans (<20%) were made. Sample size is 510. Recruitment within a year is supported by the group's prior research [more than 1000 inductions per year at IWK Grace ( the centre's name officially changed in November, 2000, to IWK Health Centre)].

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* gestational age 37 weeks or more based on ultrasound before 24 weeks
* live single fetus in cephalic presentation
* indication for induction of labour

Exclusion Criteria:

* non reassuring fetal heart rate tracing
* maternal prior uterine surgery
* known hypersensitivity to misoprostol or other prostaglandin
* contraindication to vaginal birth
* fetal anomaly identified on antenatal ultrasound
* uncontrolled maternal asthma or epilepsy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women giving birth at the IWK Health Centre
Enrollment: 511 (Actual)
Dates: Start 1999-04-01 (Actual); Primary Completion 2000-12-01 (Actual); Study Completion 2000-12-01 (Actual)

PRIMARY OUTCOMES:
Time interval from induction (at randomization) to vaginal birth | Randomization to newborn vaginal birth, assessed through to study completion, up to 10 weeks
  The chosen clinically important difference: 4 hours (240 minutes) difference. Caesarean sections could not be included in this planned parametric analysis (ANOVA) comparison of means

SECONDARY OUTCOMES:
Time interval from induction (at randomization) to birth | Randomization to newborn birth, assessed through to study completion, up to 10 weeks
  Rank order nonparametric analysis [Kruskal Wallis (KW)] where a Caesarean is a failure to deliver vaginally and ranked longer than any vaginal birth- comparison of medians (KW ANOVA).
Profound newborn acidemia | Cord blood gas sample collected at birth
  Frequency of newborns with umbilical cord blood arterial pH < 7.0
Newborn respiratory depression | Assessed at 5 minutes after birth
  Frequency of newborns with Apgar score at 5 minutes < 4
Newborn birth asphyxia | Birth to newborn hospital discharge, assessed up to 10 weeks
  Frequency of participants whose newborn experiences birth asphyxia as defined in the American College of Obstetrics and Gynecology Committee Opinion # 197 (Int J Gynecol Obstet 1998;61:309-10). The newborn with birth asphyxia must have each of the following four criteria :[1] profound academia (umbilical cord blood arterial pH< 7.0, obtained at birth); and (2) Apgar score <4 at five minutes as assessed by neonatal caregivers; and [3] neonatal neurologic sequelae (newborn with one or more of seizures, hypotonia, coma);and [4] dysfunction in one or more of the cardiovascular, gastrointestinal, hematologic, pulmonary, hepatic or renal systems. Criteria (3) and (4) are as assessed by neonatal caregivers from birth to newborn hospital discharge.
Newborn severe metabolic acidemia | Cord blood gas sample collected at birth
  Frequency of newborns with umbilical cord arterial blood base deficit >16.0 mmol/L
Newborn moderate metabolic acidemia | Cord blood gas sample collected at birth
  Frequency of newborns with umbilical cord arterial blood base deficit >12.0 mmol/L
Birth method | At newborn birth
  Frequency of spontaneous, operative vaginal (vacuum and/or forceps), or caesarean birth
Oxytocin Use | Randomization to maternal delivery, assessed through to study completion, up to 10 weeks
  Frequency of participants who received intrapartum use of oxytocin for labor augmentation or induction
Epidural Use | Randomization to maternal delivery, assessed through to study completion, up to 10 weeks
  Frequency of participants who received an epidural for intrapartum analgesia
Perineal Trauma | Randomization to maternal hospital discharge, assessed up to 10 weeks
  Frequency of participants who had received suture perineal repair of a laceration or episiotomy
Caesarean Section | At newborn birth
  Frequency of Caesarean section
Maternal nausea | Randomization to maternal delivery, assessed through to study completion, up to 10 weeks
  Frequency of participants who had nausea during labor
Maternal vomiting | Randomization to maternal delivery, assessed through to study completion, up to 10 weeks
  Frequency of participants who had vomiting during labor
Maternal diarrhea | Randomization to maternal delivery, assessed through to study completion, up to 10 weeks
  Frequency of participants experiencing diarrhea during labor
Excessive uterine activity | Randomization to birth, assessed through to study completion, up to 10 weeks
  Frequency of tachysystole and/or hyperstimulation - blind review of fetal heart rate, uterine contraction tracings by research team physician, remote from delivery.

OTHER OUTCOMES:
Vaginal birth in less than 24 hours | Randomization to newborn birth, assessed through to study completion, up to 10 weeks
  Frequency of newborns with vaginal birth in less than 24 hours from randomization (induction).
Time interval from randomization to full dilation | Randomization to newborn birth, assessed through to study completion, up to 10 weeks
  ANOVA analysis for mothers with vaginal birth
First stage of labor duration | Randomization to newborn birth, assessed through to study completion, up to 10 weeks
  ANOVA analysis of time interval from labor onset to full dilation for mothers with vaginal birth
Second stage of labor duration | Randomization to newborn birth, assessed through to study completion, up to 10 weeks
  ANOVA analysis of time interval from full dilation to vaginal birth for mothers with vaginal birth
Maternal satisfaction questionaire | Randomization to maternal hospital discharge, assessed up to 10 weeks
  ANOVA analysis of participants' total score on the Labour Agentry Scale(LAS). The LAS will be given to consenting participants as a written questionnaire prior to maternal discharge. A mother will be asked to try to remember how she felt during her recent birth experience. If a response is not received by eight weeks following maternal discharge a single reminder telephone contact will made. The LAS is a seven point Likert scale. It measures a mother's sense of control during labor. Score range is from one to seven on each of 18 items. The minimum score is 18 and maximum score is 126. A higher score indicates a greater sense of control. (Hodnett ED, Simmons-Tropea DA. The Labour Agentry Scale: Psychometric properties of an instrument measuring control during childbirth. Res Nurs Health 1987;10:301-10)
Maternal satisfaction choice | Randomization to maternal hospital discharge, assessed up to 10 weeks
  Frequency of response (yes/no) by participants to written question "If you needed a labor induction in another pregnancy would you want to have the same induction method ?" This question was administered with the questionnaire in Outcome 21 above, given to mother prior to hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: David C Young, MD MSc FRCSC, Principal Investigator — IWK Health Centre; B A Armson, MD MSc FRCSC, Study Director — IWK Health Centre

IPD SHARING:
Plan to Share IPD: No
no sharing plan is in place